CLINICAL TRIAL: NCT04480879
Title: A Randomised, 3 Period, Single Dose, Open-label Crossover Study to Evaluate the Systemic Exposure of AZD8154 While Administered Via Inhalation Using a Nebuliser Formulation and a Monodose Dry Powder Inhaler (DPI) Formulation in Healthy Subjects
Brief Title: Evaluation of AZD8154 Concentrations in Blood
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Need for evaluation of emerging pre-clinical toxicology findings
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D8900C00005
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: Phase 1, Phosphoinositide 3-kinase inhibitor, open-label crossover study
MeSH Terms: conditions — Asthma | interventions — Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AZD8154 nebuliser suspension (Experimental): The study subjects will receive 1 mg delivered dose of AZD8154 nebuliser suspension
  Interventions: Drug: AZD8154 nebuliser
- AZD8154 Monodose (Experimental): The study subjects will receive 1 mg capsule delivered dose of AZD8154 Monodose DPI formulation
  Interventions: Drug: AZD8154 Monodose DPI presented in capsules
- AZD8154 Placebo Monodose DPI (Placebo Comparator): The study subjects will receive AZD8154 placebo Monodose DPI formulation dosed to correspond to 1 mg delivered dose AZD8154 Monodose DPI formulation
  Interventions: Drug: AZD8154 Placebo Monodose DPI presented in capsules

INTERVENTIONS:
Drug: AZD8154 nebuliser — Nebuliser suspension
  Arms: AZD8154 nebuliser suspension
Drug: AZD8154 Monodose DPI presented in capsules — AZD8154 Monodose DPI formulation delivered dose
  Arms: AZD8154 Monodose
Drug: AZD8154 Placebo Monodose DPI presented in capsules — The dose correspond to AZD8154 Monodose DPI formulation
  Arms: AZD8154 Placebo Monodose DPI

SUMMARY:
This study is intended to evaluate the systemic pharmacokinetic (PK) characteristics and the safety of AZD8154 following administration of the Monodose DPI formulation compared with the administration of the nebuliser suspension.

DETAILED DESCRIPTION:
This study will be a randomised, open-label, 3-period, single-dose, single-centre, crossover study in healthy males and healthy females of non-childbearing potential.

The study will comprise:

* A Screening Period of maximum 28 days;
* Three treatment periods during which subjects will be resident at the Clinical Unit from the morning of the day before dosing with AZD8154 or placebo (Day 1) until 72 hours following dosing for collection of PK samples; discharged on the morning of Day 4 of each treatment period;
* A Follow up Visit within 6 ± 1 days after last dose administration of investigational medicinal products (IMPs) (i.e., AZD8154 or placebo).

A total of 15 healthy subjects will be randomised in this study to ensure that at least 12 subjects are evaluable.

Each subject will be involved in the study for approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or healthy female subjects of non childbearing potential aged 18 to 55 years (inclusive at the Screening Visit) with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at Screening Visit and on admission to the Clinical Unit, must not be lactating and must be of non childbearing potential, confirmed at Screening by fulfilling 1 of the following criteria (i) Females are considered postmenopausal if they have had amenorrhea for at least 12 months without an alternative medical cause. The following age specific requirements apply: Women under 50 years old are considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments and with luteinising hormone and follicle stimulating hormone levels are in the postmenopausal range.

   Women over 50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments.

   (ii) Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 60 kg and no more than 100 kg inclusive.
5. Subject has a forced expiratory volume in 1 second ≥ 80% of the predicted value regarding age, height, gender and ethnicity at the Screening Visit.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Principal Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. Subject is immune compromised.
3. History of diabetes, impaired fasting glucose, metabolic syndrome, hypertriglyceridemia or familial lipid disorders.
4. Current or previous history of malignancy of any kind except cutaneous basal or squamous cell carcinoma successful treated with therapy.
5. History of any respiratory disorders such as asthma, chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis (IPF), or infantile bronchiolitis.
6. Subject with latent or active tuberculosis, as confirmed by a positive QuantiFERON® TB Gold test or as judged by the Investigator at the Screening Visit.
7. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs, or bowel disorders not otherwise specified.
8. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the IMP.
9. Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results, defined as the following:

   (i) Alanine aminotransferase and/or aspartate aminotransferase > 1.5 x the upper limit of the normal (ULN) laboratory range.

   (ii) Bilirubin > 1.5 times the ULN laboratory range. (iii) Absolute neutrophil count < lower limit of normal (LLN). (iv) Absolute lymphocyte count < LLN.
10. Any positive result at the Screening Visit for serum hepatitis B surface antigen OR hepatitis B core antibodies, hepatitis C virus antibody (anti HCV) and human immunodeficiency virus.
11. Abnormal vital signs, after 5 minutes supine rest, defined as any of the following:

    (i) Systolic blood pressure (BP) < 90 mmHg or > 140 mmHg. (ii) Diastolic BP < 50 mmHg or > 90 mmHg. (iii) Pulse < 50 or > 90 beats per minute (bpm).
12. Any clinically important abnormalities in rhythm, conduction or morphology of the 12 lead safety ECG as judged by the Investigator.

    (i) Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome.

    (ii) PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre excitation).

    (iii) PR (PQ) interval prolongation (> 220 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation.

    (iv) Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g., ventricular hypertrophy or pre excitation.
13. Previous use of a mechanistic target of rapamycin (mTOR) antagonist (e.g., rapamycin, everolimus) or PI3K inhibitor (selective or non selective PI3K inhibitors).
14. Known or suspected history of drug abuse as judged by the Investigator.
15. Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the previous 3 months.
16. History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.
17. Positive screen for drugs of abuse or cotinine (nicotine) at the Screening Visit or admission to the Clinical Unit or positive screen for alcohol on admission to the Clinical Unit before the first administration of the IMP.
18. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD8154.
19. Receipt of live attenuated vaccines 2 months before first administration of the IMP and 3 months after the last IMP administration.
20. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the Investigator.
21. Use of drugs with cytochrome P450 (CYP) 3A enzyme inducing or inhibition properties within 3 weeks before first administration of IMP.
22. Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks before the first administration of the IMP or longer if the medication has a long half life.
23. Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss > 500 mL during the 2 months before the Screening Visit.
24. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration the IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.
25. Involvement of any Astra Zeneca or study site employee or their close relatives.
26. Judgement by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
27. Subjects who cannot communicate reliably with the Investigator and/or is not able to read speak and understand the German language.
28. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship or committed to an institution by governmental or juridical order.
29. Subject has a positive test result for SARS-CoV-2 RT-PCR before randomisation.
30. Subject has clinical signs and symptoms consistent with COVID-19, e.g., fever, dry cough, dyspnoea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on first admission.
31. History of severe COVID-19 (hospitalisation, extracorporeal membrane oxygenation, mechanically ventilated).
32. Subjects who are regularly exposed to COVID-19 as part of their daily life (e.g., health care professionals working in COVID-19 wards or at emergency departments).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve from zero to infinity (AUCinf) | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate the PK characteristics of AZD8154 following inhaled single dose administration of a Monodose DPI formulation when compared with inhaled single dose administration of a nebuliser suspension.
Area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUClast) | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate the PK characteristics of AZD8154 following inhaled single dose administration of a Monodose DPI formulation when compared with inhaled single dose administration of a nebuliser suspension.
Maximum observed plasma (peak) drug concentration (Cmax) | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate the PK characteristics of AZD8154 following inhaled single dose administration of a Monodose DPI formulation when compared with inhaled single dose administration of a nebuliser suspension.
Dose normalised AUCinf | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate the PK characteristics of AZD8154 following inhaled single dose administration of a Monodose DPI formulation when compared with inhaled single dose administration of a nebuliser suspension.
Dose normalised AUClast | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate the PK characteristics of AZD8154 following inhaled single dose administration of a Monodose DPI formulation when compared with inhaled single dose administration of a nebuliser suspension.
Dose normalised Cmax | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate the PK characteristics of AZD8154 following inhaled single dose administration of a Monodose DPI formulation when compared with inhaled single dose administration of a nebuliser suspension.

SECONDARY OUTCOMES:
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate further PK parameters of AZD8154 following inhaled single dose administration of a Monodose DPI formulation and an inhaled single dose administration of a nebuliser suspension.
Half life associated with terminal slope of a semi logarithmic concentration time curve (t½λz) | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate further PK parameters of AZD8154 following inhaled single dose administration of a Monodose DPI formulation and an inhaled single dose administration of a nebuliser suspension.
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRT) | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate further PK parameters of AZD8154 following inhaled single dose administration of a Monodose DPI formulation and an inhaled single dose administration of a nebuliser suspension.
Terminal elimination rate constant (λz) | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate further PK parameters of AZD8154 following inhaled single dose administration of a Monodose DPI formulation and an inhaled single dose administration of a nebuliser suspension.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate further PK parameters of AZD8154 following inhaled single dose administration of a Monodose DPI formulation and an inhaled single dose administration of a nebuliser suspension.
Volume of distribution following extravascular administration (based on terminal phase) (Vz/F) | Study Day 1 to 4 (Pre dose, 10 minutes, 30 minutes, 45 minutes, 1, 2, 3, 4, 6, 12, 18, 24, 36, 48 and 72 hours post dose)
  To evaluate further PK parameters of AZD8154 following inhaled single dose administration of a Monodose DPI formulation and an inhaled single dose administration of a nebuliser suspension.
Number of subjects with adverse events | Day-1, 1 to 4 (Spontaneous plus pre dose, 3, 12, 24, 48 and 72 hrs post dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal blood pressure | At screening (Day-28 to-2), Day-1, Day1 to 4 (Predose and 72hrs post dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal pulse rate | At screening (Day-28 to-2), Day-1, Day1 to 4 (Predose and 72hrs post dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal tympanic temperature | At screening (Day-28 to-2), Day-1, Day 1 to 4 (Predose, 24, 48, and 72 hrs post dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal respiratory rate | At screening (Day-28 to-2), Day-1, Day1 to 4 (Predose and 72hrs post dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal ECG | At screening (Day-28 to-2), Day-1, Day 1 to 4 (Predose and 72 hrs post dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal physical examination | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal spirometry | At screening(Day-28 to-2), Day-1, Day1 to 4 (Predose and 30min, 90min, 3hrs, 12hrs and 24hrs postdose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal White blood cell (WBC) count | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Red blood cell (RBC) count | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Haemoglobin (Hb) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Haematocrit (HCT) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Mean corpuscular volume (MCV) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Mean corpuscular haemoglobin (MCH) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Mean corpuscular haemoglobin concentration (MCHC) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Neutrophils absolute count | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Lymphocytes absolute count | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Monocytes absolute count | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Eosinophils absolute count | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Basophils absolute count | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Platelets | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Reticulocytes absolute count | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Sodium | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Potassium | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Urea | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Creatinine | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Albumin | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Calcium | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Phosphate | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Glucose(fasting) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal C-reactive protein (CRP) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Alkaline phosphatase (ALP) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Alanine aminotransferase (ALT) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Aspartate aminotransferase (AST) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Gamma glutamyl transpeptidase (GGT) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Total Bilirubin (TBL) | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Unconjugated bilirubin | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects
Number of subjects with abnormal Urinalysis | At screening (Day-28 to-2), Day-1, Day1 to 4 and follow-up visit (6± 1 days post last dose)
  To assess the safety of single doses of AZD8154 (Monodose DPI formulation and nebuliser suspension) or placebo (Monodose DPI formulation) in healthy subjects.
  The parameters to be assessed are glucose, protein and blood in urine

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home